CLINICAL TRIAL: NCT00837070
Title: Percutaneous Rupture of Zygapophyseal Joint Cysts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Principal Investigator, Therese Seierstad, Head of Research, Division for Radiology and Nuclear Medicine, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 264-07111a 2007.345
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Zygapophyseal Synovial Joint Cyst
Keywords: Zygapophyseal; joint; cyst; Fluoroscopy; guided; percutaneous; Lumbar
MeSH Terms: conditions — Cysts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Percutaneous zygapophyseal cyst rupture
  Interventions: Procedure: Percutaneous zygapophyseal cyst rupture

INTERVENTIONS:
Procedure: Percutaneous zygapophyseal cyst rupture — Patients will be treated by introducing a 20G spinal needle in the inferior joint recess of the zygapophyseal joint.1 ml of celestone-chronodose,1 ml of Marcain 5 mg/ml and 1-3 ml of contrast media:Omnipaque 240 will be injected until the cyst ruptures.
  Other Names: Axiom Artis Siemens

SUMMARY:
Lumbar zygapophyseal joint cysts can cause lower extremity radiculopathy. These cysts can be cured by a minimally invasive technique: percutaneous cyst distention and rupture

DETAILED DESCRIPTION:
Lumbar zygapophyseal joint cysts can cause lower extremity radiculopathy. These cysts can be cured by a minimally invasive technique: percutaneous cyst distention and rupture.

30 patient with lower extremity radiculopathy caused by lumbar zygapophyseal joint cysts will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lumbar zygapophyseal joint cyst and compression of a spinal nerve root with lower extremity radiculopathy proven by MRI.

Exclusion Criteria:

* Infection, uncontrollable bleeding disorder

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
VAS(Visual analogue scale)for extremity pain | 1-3 and 12 months after intervention

SECONDARY OUTCOMES:
Roland-Morris disability index | 1-3 and 12 months after intervention
Reduction of cyst size based om T2 MRI | 3 and 12 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Øivind Gjertsen, Md, Msc, Principal Investigator — Oslo University Hospital
Locations (1):
- Departement of Neuroradiology Oslo university hospital avd Ullevaal, Oslo, Norway